CLINICAL TRIAL: NCT01774630
Title: Multicenter Single-arm Pilot Study Evaluating Efficacy of Nilotinib in CML Patients With Molecular Relapse After Glivec Discontinuation Within the Context of the STIM Trials (STIM and STIM2)
Acronym: NiloPost-STIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2012/18
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive
Keywords: Treatment, relapse, complete molecular response
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Recurrence | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nilotinib (Experimental): 300 mg/twice a day
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — 300 mg/twice a day

SUMMARY:
Chronic myeloid leukemia (CML) is a hematopoietic neoplasm characterized by the reciprocal translocation t(9;22). The resulting oncoprotein, bcr-abl is an essential trigger for growth and survival of leukemic cells. In the past decade, the bcr-abl tyrosine kinase inhibitor (TKI) imatinib (IM or Glivec©) has been the standard of care for patients with CML, inducing durable responses. However, requiring continuing IM indefinitely and the ability of IM to eradicate the CML clone was uncertain.

In a small proportion of patients, IM can induce complete molecular response (CMR) defined by the disappearance of the bcr-abl transcript in conventional quantitative RT-PCR. The question whether or not these patients are cured and can discontinue drug therapy has been assessed by Mahon and coll, in the STIM study. He demonstrates that IM can be safely discontinued in patient with a CMR of at least 2 year duration and all patients who relapsed after IM discontinuation mainly did it in the first 6 months and responded to reintroduction of imatinib.

Nilotinib is a rationally designed second generation tyrosine kinase inhibitor with improved target specificity over imatinib. Its efficacy and safety in the treatment of patients who are resistant or intolerant to imatinib as well as patients with newly diagnosed CML-CP led to the registration in second and first line treatment of CML-CP patients. Nilotinib produces even faster and deeper responses with more occurrence of CMR than does Imatinib. Consequently, one can assume that a more potent drug such nilotinib could induce deeper and sustained CMR allowing longer period off treatment than IM.

The objective of this pilot trial is to assess if Nilotinib can rescue STIM patients in molecular relapse after IM discontinuation and to provide an estimation about duration of CMR after nilotinib discontinuation in 2nd line therapy among patients experiencing 2 years of stable CMR with nilotinib.

DETAILED DESCRIPTION:
Patients with CML included in STIM trials, stopped their treatment by imatinib because the signal was not detectable. In case of reappearance of this transcript Bcr-Abl, the patient relapses. The trial Nilo Post STIM is suggested to the patient to assess if Nilotinib can rescue STIM patients in molecular relapse after IM discontinuation and to provide an estimation about duration of CMR after nilotinib discontinuation in 2nd line therapy among patients experiencing 2 years of stable CMR with nilotinib.

The treatment/strategy for this study:

* Screening

  * Inclusion/exclusion criteria
  * CML history
  * Confirm molecular relapse after discontinuation of imatinib (quantitative RT-PCR on two consecutive assessments from peripheral blood samples)
* Treatment

  • Nilotinib 300mg BID for 2 years
  * Premature treatment discontinuation while on study: primary or secondary resistance progression to accelerated phase or blast crisis, AE (to be defined later).
  * In case of unsatisfactory response: transcript stability or increase on two consecutive PCR: nilotinib blood monitoring, and nilotinib dose escalation up to 400mg BID will be proposed
  * Discontinuation at 2 years for patients who resumed confirmed CMR
* Follow-up while on treatment with nilotinib:

  * Physical exam, basic laboratory parameters, monthly during the first 3 months then every 3 months.
  * Centralized quantitative RT-PCR for Bcr-Abl monthly for 6 months then every 3 months for 24 months
  * Follow AE management guidelines for nilotinib reduction/interruptions
* Follow-up after nilotinib discontinuation

  * Patients in confirmed molecular relapse

    * Physical exam, event collection, basic laboratory parameters (including glycemic and lipid profile) every 2 months during the first year then every 3 months
    * Hematology and centralized quantitative RT-PCR monthly the first year then every 3 months for 12 months
  * Patients without confirmed molecular relapse will take another treatment (dasatinib for example) and will stop their follow-up in the trial

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Patient participating to the STIM trials (including STIM, STIM2 et EURO-SKI) and with confirmed molecular relapse on two consecutive RQ PCR, after imatinib discontinuation
* Still in chronic phase
* Not yet treated for this relapse
* At least 18 years old (no upper age limit)
* SGOT and SGPT < 2.5 UNL
* Serum creatinin < 2 UNL
* No planned allogeneic stem cell transplantation
* Signed informed consent
* ECOG score 0 to 2

Exclusion Criteria:

* Pregnancy, lactation
* Prior or concurrent malignancy other than CML (exceptions to be mentioned)
* Serious uncontrolled cardiovascular disease
* Severe psychiatric/neurological disease (previous or ongoing)
* Ongoing treatment at risk for inducing "torsades de pointe"
* QTcF > 450ms despite correction of predisposing factors (i.e electrolytes…)
* Congenital long QTcF
* No health insurance coverage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-04-10 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Estimated survival rate of patients without molecular relapse 3 years after enrollment | Evaluation by RTq-PCR monthly the first year of treatment with nilotinib then every 3 months until 24 months, date of discontinuation of Nilotinib for patients in sustained complete molecular response (CMR). After discontinuation of Nilotinib patie
  CMR is defined as >5 log reduction in Bcr-Abl and Abl levels and undetectable transcripts on quantitative RTq-PCR

SECONDARY OUTCOMES:
Rate and kinetics of CMR while on treatment with nilotinib | at 6 and 12 months of treatment with nilotinib
  Same definition of CMR as above
Duration of CMR while on treatment with nilotinib | Any time
  Defined as the time from the date of first documented CMR to the date of first confirmed molecular relapse defined as positivity of Bcr-Abl transcripts in quantitative RT-PCR with a ratio of bcr-abl to Abl ≥ 10-5, as confirmed by a second analysis point at two successive assessments
Event free survival (EFS) | Any time
  Events include loss of major molecular response (MMR) , loss of complete cytogenetic response (CCyR) loss of complete hematologic response (CHR), progression to accelerated phase and blst crisis (AP-BC), death whatever the cause, adverse-event leading to premature discontinuation of nilotinib
Safety tolerability of nilotinib and compliance | Any time
  Haematological and non-haematological adverse events (AE) graded will be according to the NCI CTC AE v4. Compliance will be estimated using the 4 items Morisky scale
Duration of CMR after nilotinib discontinuation | Measured from the start of nilotinib discontinuation to the date of first confirmed molecular relapse as defined above
Event free survival (EFS) | Overall and after nilotinib discontinuation
  Same events as for EFS described above
Predictive factors of maintained CMR after nilotinib discontinuation: sex, Sokal risk score at diagnosis, duration of previous treatment with imatinib, CMR duration before and after discontinuation of imatinib | After discontinuation of nilotinib
  Parameters will be recorded before and after both sequences of treatment imatinib and nilotinib

CONTACTS AND LOCATIONS:
Overall Officials: Viviane DUBRUILLE, Study Chair — Nantes University Hospital; Gabriel ETIENNE, Study Chair — University Hospital Bordeaux, France; Franck NICOLINI, Study Chair — Hospices Civils de Lyon; Delphine REA, Study Chair — APHP, St Louis Hospital
Locations (10):
- France (10):
  - CHU Angers, Angers
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier de Versailles - Hôpital André Mignot - Service de Médecine B, Le Chesnay
  - CHU de Nice, Service Hématologie Clinique, Nice
  - Hôpital Haut Lévêque, Service Hématologie, Pessac
  - Centre Hospitalier Lyon Sud, Service Hématologie, Pierre-Bénite
  - CH d'Annecy, Pringy
  - Hôpital Pontchaillou, Rennes
  - CHU de Toulouse, Service d'Hématologie, Toulouse
  - CH Valence, Valence

IPD SHARING:
Plan to Share IPD: No